CLINICAL TRIAL: NCT03571724
Title: A Longitudinal Ambulatory Study to Assess Changes in Cigarette Consumption and Biomarkers of Exposure During a 6-week Switch to Very Low Nicotine Cigarettes
Brief Title: A Study to Assess Changes in Cigarette Consumption During a Switch to Very Low Nicotine Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 22nd Century Group, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CA24914
Record Dates: First submitted 2018-06-02; First posted 2018-06-28 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Tobacco Use
Keywords: Very Low Nicotine; Cigarette; VLN
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: Longitudinal ambulatory switching study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Brand (UB) non-mentholated filtered cigarettes (Experimental): Usual Brand (UB) mentholated filtered cigarettes Usual Brand (UB) non-mentholated filtered cigarettes or to very low nicotine non-mentholated cigarettes
  Interventions: Other: Non-Menthol Very Low Nicotine Cigarettes; Other: Subject's UB non-mentholated filtered cigarettes
- Usual Brand (UB) mentholated filtered cigarettes (Experimental): Subjects will be randomized to continue to smoke Usual Brand (UB) mentholated filtered cigarettes or to very low nicotine mentholated cigarettes
  Interventions: Other: Menthol Very Low Nicotine Cigarettes; Other: Subject's UB mentholated filtered cigarettes

INTERVENTIONS:
Other: Non-Menthol Very Low Nicotine Cigarettes — King size non-menthol cigarettes containing 0.4mg nicotine /g tobacco
  Arms: Usual Brand (UB) non-mentholated filtered cigarettes
Other: Menthol Very Low Nicotine Cigarettes — King size menthol cigarettes containing 0.4mg nicotine /g tobacco
  Arms: Usual Brand (UB) mentholated filtered cigarettes
Other: Subject's UB non-mentholated filtered cigarettes — King size non-menthol cigarettes
  Arms: Usual Brand (UB) non-mentholated filtered cigarettes
Other: Subject's UB mentholated filtered cigarettes — King size menthol cigarettes
  Arms: Usual Brand (UB) mentholated filtered cigarettes

SUMMARY:
This study evaluates the impact of switching from usual brand cigarettes to very low nicotine cigarettes on cigarette consumption, smoking behavior, and biomarkers of exposure.

DETAILED DESCRIPTION:
Very low nicotine (VLN) cigarettes contain a 'non-additive' level of nicotine. This study will switch smokers from their usual brand to VLN cigarettes. Periodically during the study the investigators will collect blood and measure nicotine exposure and also other biomarkers to see what effect switching has. The participants will also use a diary to record number of cigarettes smoked. Cigarette butts will also be collected.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study.

1. Is a healthy adult male or female adult smoker, 26 to 65 years of age, inclusive, at Screening.
2. Has been a smoker for at least 5 years prior to Screening. Brief periods of non smoking (e.g., up to 7 consecutive days due to illness, trying to quit, participation in a study where smoking was prohibited) during that time will be permitted at the discretion of the Investigator.
3. Reports smoking an average of 10 or more manufactured combustible cigarettes per day at Screening.
4. Usual brand (UB) of cigarette is a filtered king size cigarette (with an approximate length of 84 mm (± 3 mm)).
5. Has a positive urine cotinine (≥ 500 ng/ml) at Screening.
6. Has an exhaled Carbon Monoxide > 10 ppm at Screening.
7. If female, has a negative serum pregnancy test at Screening.
8. A female subject of childbearing potential must have been using one of the following forms of contraception and agree to continue using it through completion of the study:

   * hormonal (e.g., oral, vaginal ring, transdermal patch, implant, or injection) consistently for at least 3 months prior to Screening;
   * double barrier method (e.g., condom with spermicide, diaphragm with spermicide) consistently for at least 14 days prior to Screening;
   * intrauterine device for at least 3 months prior to Screening;
   * Essure® or similar nonsurgical sterilization procedure at least 6 months prior to Screening
   * a partner who has been vasectomized for at least 6 months prior to Screening;
   * abstinence beginning at least 14 days prior to Screening and through the End of Study.
9. A female subject of non childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to Screening:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; Or be postmenopausal with amenorrhea for at least 1 year prior to Day 1 and follicle stimulating hormone (FSH) levels consistent with postmenopausal status.
10. Willing to comply with the requirements of the study, including a willingness to use the test products.
11. Voluntary consent to participate in this study documented on the signed informed consent form (ICF).
12. Subject is not planning to leave the area during the course of the study.

Exclusion Criteria:

Subjects may be excluded from the study if there is evidence of any of the following criteria at Screening, start of Week -1 (first clinic visit), or during the study as noted, in the opinion of the Investigator.

1. History or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary (especially bronchospastic diseases and asthma), immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Clinically significant abnormal findings on the physical examination, medical history, ECG, or clinical laboratory results, in the opinion of the Investigator.
3. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
4. An acute illness (e.g., upper respiratory infection, viral infection) requiring treatment with prescription medication(s) within 14 days prior to Screening or first clinic visit.
5. Fever (>100.5 degrees F) at Screening or first clinic visit.
6. Body mass index (BMI) greater than 40.0 kg/m2 or less than 18.0 kg/m2 at Screening.
7. History of drug or alcohol abuse or has used medical/recreational marijuana within 12 months of Screening.
8. Diabetes mellitus that is not controlled by diet/exercise alone, in the opinion of the Investigator.
9. Seated heart rate is lower than 40 bpm or higher than 99 bpm at Screening, unless deemed not clinically significant by the PI.
10. Seated systolic blood pressure <90 mmHg or >150 mmHg, diastolic blood pressure <40 mmHg or >95 mmHg at Screening, unless deemed not clinically significant by the PI.
11. Positive urine screen for drugs of abuse or alcohol at Screening or at the first clinic visit.
12. Female subjects who are pregnant, lactating, or intend to become pregnant from Screening through the End of Study.
13. Use of medications known to interact with cytochrome p450 2A6 (including, but not limited to, amiodarone, desipramine, isoniazid, ketoconazole, miconazole, phenobarbital, rifampin, tranylcypromine, methoxsalen) within 3 months prior to Screening and throughout the study.
14. Use of inhalers to treat any medical condition within 3 months prior to Screening and throughout the study.
15. Use of nicotine-containing products other than factory manufactured cigarettes [e.g., roll-your-own cigarettes, e-vapor products, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum] within 28 days prior to Screening.
16. Use of any prescription smoking cessation treatments, including, but not limited to, varenicline (Chantix®) or buproprion (Zyban®) within 3 months prior to Screening.
17. Self-reported puffer/non-inhaler (i.e., a smoker who draws smoke from the cigarette into the mouth and throat but does not inhale).
18. Planning to quit smoking during the study period or postponing a quit attempt in order to participate in the study.
19. Plasma donation within 7 days prior to Screening or at any time during the study.
20. Donation of blood or blood products (with the exception of plasma as noted above), had significant blood loss, or received whole blood or a blood product transfusion within 56 days prior to Screening.
21. Participation in a previous clinical study for an investigational drug, device, biologic, or tobacco product within 30 days prior to Screening.
22. Subject or a first-degree relative (i.e., parent, sibling, child) is a current or former employee of the tobacco industry or a named party or class representative in litigation with the tobacco industry.
23. Subject or a first-degree relative (i.e., parent, sibling, child) is a current employee of the clinic sites.

Ages: 26 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L Matthew, MD, Principal Investigator — Celerion; Melanie Fein, Principal Investigator — High Point Clinical Trials
Locations (2):
- United States (2):
  - Celerion, Lincoln, Nebraska
  - High Point Clinical Trials, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 142 smokers were recruited from two sites in the United States; Celerion, Lincoln Nebraska and High Point Clinical Trials Center, High Point, North Carolina. The participants were recruited via social media, print, TV, radio, referrals.
Pre-assignment Details: Subjects may have been excluded from the study if there was evidence of any of the exclusion criteria during the study as noted, in the opinion of the Investigator.
Groups:
- Non-Menthol Very Low Nicotine Cigarettes: Subjects will be switched from their usual brand to smoke Very Low Nicotine king size cigarettes
  Non-Menthol Very Low Nicotine Cigarettes: King size non-menthol cigarettes containing 0.4mg nicotine /g tobacco
- Menthol Very Low Nicotine Cigarettes: Subjects will be switched from their usual brand to smoke Very Low Nicotine king size Menthol cigarettes
  Menthol Very Low Nicotine Cigarettes: King size menthol cigarettes containing 0.4mg nicotine /g tobacco
- Usual Brand Non-Metholated: Subjects continue to smoke their usual brand non-Menthol cigarettes
- Usual Brand Metholated: Subjects continue to smoke their usual brand Menthol cigarettes
Period: Week -1 (Prior to Switching)
Arm/Group | Non-Menthol Very Low Nicotine Cigarettes | Menthol Very Low Nicotine Cigarettes | Usual Brand Non-Metholated | Usual Brand Metholated
Started | 0 | 0 | 72 | 70
Topography | 0 | 0 | 18 (These subjects switched into VLN arms.) | 18 (These subjects switched into VLN arms.)
PK Nicotine | 0 | 0 | 12 (These subjects switched into VLN arms.) | 12 (These subjects switched into VLN arms.)
Completed | 0 | 0 | 72 | 70
Not Completed | 0 | 0 | 0 | 0
Period: Week 1-6
Arm/Group | Non-Menthol Very Low Nicotine Cigarettes | Menthol Very Low Nicotine Cigarettes | Usual Brand Non-Metholated | Usual Brand Metholated
Started | 50 (Non-menthol VLN subjects were assigned to this arm after randomization at week 1) | 50 (Menthol VLN subjects were assigned to this arm after randomization at week 1) | 22 | 20
Completed | 43 | 42 | 19 | 20
Not Completed | 7 | 8 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Brand Non-Mentholated: Subjects will continue to use their usual brand non-menthol cigarettes
- Usual Brand Mentholated: Subjects will continue to use their usual brand menthol cigarettes
- Total: Total of all reporting groups
Arm/Group | Non-Menthol Very Low Nicotine Cigarettes | Menthol Very Low Nicotine Cigarettes | Usual Brand Non-Mentholated | Usual Brand Mentholated | Total
Number analyzed (Participants) | 50 | 50 | 22 | 20 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (10.85) | 40.5 (9.34) | 45.8 (12.39) | 42.7 (10.82) | 43.5 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 9 | 10 | 60
  Male | 31 | 28 | 13 | 10 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 49 | 49 | 21 | 19 | 138
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 29 | 2 | 12 | 46
  White | 44 | 17 | 18 | 8 | 87
  More than one race | 1 | 2 | 1 | 0 | 4
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 22 | 20 | 142
Cigarettes Per Day (CPD) [Mean (Standard Deviation); unit: Cigarettes per day] — Smoking history summary (safety, ITT population) for cigarettes per day for the VLN non-mentholated, VLN mentholated, UB non-mentholated and UB mentholated.
  Cigarettes per day | 19.8 (6.92) | 15.4 (6.19) | 18.2 (3.85) | 17.1 (6.16) | 17.6 (6.39)

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Per Day
Description: Primary objective is to measure a change in cigarette consumption behavior before, during and after switching from usual brand to to VLN cigarettes. Subjects will record their cigarette consumption daily in an electronic diary. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).All 142 randomized subjects were included in the ITT population based on product use. Out of these, 71 subjects were included in the PP Population and 71 were excluded. All excluded subjects had a ratio of [plasma cotinine/CPD VLN]/[plasma cotinine/CPD baseline] > 0.2. It was pre-specified to exclude participants with a ratio >0.2 as they were considered non-compliant.
Time Frame: Assessed daily from Week -1 to Week 6; Week -1, Week 2, and Week 6 reported
Population: Cigarettes per Day were calculated as the average cigarettes smoked per day in each week.
Measure: Mean (Standard Deviation); unit: Cigarettes Per Day (CPD)
Groups:
- Very Low Nicotine Mentholated; Very Low Nicotine Non-Mentholated; Very Low Nicotine Combined; Usual Brand Mentholated; Usual Brand Non-Mentholated; Usual Brand Combined: Subjects were randomized to one of four study product groups, with menthol cigarette smokers randomized to either their usual brand menthol cigarettes or VLN mentholated cigarettes, and non-menthol cigarette smokers randomized to their usual brand non-menthol cigarettes or VLN non-mentholated cigarettes.
Arm/Group | Very Low Nicotine Mentholated | Very Low Nicotine Non-Mentholated | Very Low Nicotine Combined | Usual Brand Mentholated | Usual Brand Non-Mentholated | Usual Brand Combined
Number analyzed (Participants) | 17 | 12 | 29 | 20 | 22 | 42
Cigarettes Per Day (CPD)
  Week -1 | 14.75 (6.198) | 17.19 (4.727) | 15.76 (5.676) | 16.29 (5.809) | 16.80 (4.015) | 16.55 (4.895)
  Week 2: number analyzed (Participants) | 15 | 11 | 26 | 20 | 22 | 42
  Week 2 | 15.66 (7.860) | 23.32 (9.717) | 18.90 (9.341) | 15.47 (4.425) | 16.17 (4.475) | 15.84 (4.411)
  Week 6: number analyzed (Participants) | 10 | 11 | 21 | 20 | 20 | 40
  Week 6 | 14.43 (9.435) | 21.20 (8.219) | 17.98 (9.265) | 14.69 (4.877) | 15.89 (5.356) | 15.29 (5.092)

2. Secondary Outcome: Biomarkers of Exposure - Total 4-(Methylnitrosamino)-1-(3-pyridyl)-1 Butanol (NNAL)
Description: Total 24 hour urine will be collected to evaluate changes in NNAL (4-methylnitrosamino)-1-3-pyridyl)-1-butanone biomarker) before, during, and after switching to VLN cigarettes. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: Summary of Urinary NNAL Mass Excreted (ng/24 hour) by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: ng/24 hour
Groups:
- VLN Non-Mentholated; VLN Mentholated; VLN Combined; UB Non-Mentholated; UB Mentholated; UB Combined: Subjects were randomized to one of four study product groups, with menthol cigarette smokers randomized to either their usual brand menthol cigarettes or VLN mentholated cigarettes, and non-menthol cigarette smokers randomized to their usual brand non-menthol cigarettes or VLN non-mentholated cigarettes.
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 21 | 20 | 41
ng/24 hour
  Week -1 | 582.855 (288.3650) | 423.752 (185.6953) | 502.500 (253.6974) | 614.06 (353.9198) | 479.979 (203.2470) | 548.658 (294.7134)
  Week 2: number analyzed (Participants) | 48 | 43 | 91 | 21 | 20 | 41
  Week 2 | 313.911 (176.1390) | 214.139 (131.4077) | 266.766 (163.6124) | 581.039 (312.7864) | 458.036 (203.4045) | 521.037 (269.1556)
  Week 6: number analyzed (Participants) | 42 | 41 | 83 | 17 | 19 | 36
  Week 6 | 377.057 (217.6683) | 240.970 (173.1282) | 309.833 (207.3562) | 614.717 (416.6105) | 431.458 (173.9915) | 517.997 (321.7481)

3. Secondary Outcome: Biomarkers of Exposure - Total N-Nitrosonornicotine (NNN)
Description: Total 24 hour urine will be collected to evaluate changes in NNN before, during, and after switching to VLN cigarettes. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: Summary of Urinary NNAL Mass Excreted (ng/24 hour) by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: ng/24 hour
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 21 | 20 | 41
ng/24 hour
  Week -1 | 20.070 (14.4934) | 12.370 (7.9412) | 16.181 (12.2224) | 22.614 (24.4627) | 13.641 (11.1026) | 18.237 (19.4522)
  Week 2: number analyzed (Participants) | 48 | 43 | 91 | 21 | 20 | 41
  Week 2 | 14.246 (11.6548) | 9.052 (10.2762) | 11.792 (11.2701) | 20.809 (21.2301) | 12.024 (9.0103) | 16.523 (16.8430)
  Week 6: number analyzed (Participants) | 42 | 41 | 83 | 17 | 19 | 36
  Week 6 | 14.803 (11.4754) | 6.382 (4.5544) | 10.643 (9.6904) | 22.095 (25.7769) | 9.359 (6.0602) | 15.373 (19.0844)

4. Secondary Outcome: Biomarkers of Exposure - S-phenylmercapturic Acid (S-PMA)
Description: Total 24 hour urine will be collected to evaluate changes in S-PMA (benzene biomarker) before, during, and after switching to VLN cigarettes. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: Summary of Urinary S-PMA Mass Excreted (µg/24 hour) by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: µg/24 hour
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 21 | 20 | 41
µg/24 hour
  Week -1 | 7.144 (5.9255) | 6.561 (3.8833) | 6.850 (4.9823) | 7.935 (3.8120) | 8.239 (7.3290) | 8.083 (5.7274)
  Week 2: number analyzed (Participants) | 48 | 43 | 91 | 21 | 20 | 41
  Week 2 | 8.160 (7.8142) | 6.734 (4.7617) | 7.486 (6.5560) | 7.561 (3.7582) | 7.731 (5.9223) | 7.644 (4.8713)
  Week 6: number analyzed (Participants) | 42 | 41 | 83 | 17 | 19 | 36
  Week 6 | 7.282 (6.4350) | 5.589 (3.6334) | 6.446 (5.2792) | 7.261 (4.4329) | 6.845 (5.2829) | 7.042 (4.8353)

5. Secondary Outcome: Biomarkers of Exposure - 3-hydroxypropylmercapturic Acid (3-HPMA)
Description: Total 24 hour urine will be collected to evaluate changes in 3-HPMA (acrolein biomarker) before, during, and after switching to VLN cigarettes. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: Summary of Urinary 3-HPMA Mass Excreted (µg/24 hour) by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: µg/24 hour
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 21 | 20 | 41
µg/24 hour
  Week -1 | 1795.719 (708.6089) | 1644.113 (500.1249) | 1719.151 (613.8453) | 1910.675 (772.7715) | 1520.921 (605.2480) | 1720.551 (715.1892)
  Week 2: number analyzed (Participants) | 48 | 43 | 91 | 21 | 20 | 41
  Week 2 | 1706.862 (901.3990) | 1204.530 (543.2655) | 1469.496 (790.9739) | 1710.747 (732.7759) | 1329.844 (319.7909) | 1524.940 (595.1580)
  Week 6: number analyzed (Participants) | 42 | 41 | 83 | 17 | 19 | 36
  Week 6 | 1481.693 (694.6765) | 1035.064 (475.3512) | 1261.069 (634.0203) | 1815.382 (828.3606) | 1336.103 (297.2953) | 1562.429 (673.6060)

6. Secondary Outcome: Biomarkers of Exposure - 1-hydroxy Pyrene(1-OHP)
Description: Total 24 hour urine will be collected to evaluate changes in 1-OHP before, during, and after switching to VLN cigarettes. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: Summary of Urinary 1-OHP Mass Excreted (ng/24 hour) by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: ng/24 hour
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 21 | 20 | 41
ng/24 hour
  Week -1 | 334.920 (167.7463) | 315.203 (160.6678) | 324.962 (163.6689) | 314.736 (90.9545) | 316.566 (140.5579) | 315.629 (116.2823)
  Week 2: number analyzed (Participants) | 48 | 43 | 91 | 21 | 20 | 41
  Week 2 | 262.756 (157.8692) | 214.010 (117.020) | 239.722 (141.4377) | 289.071 (97.7694) | 263.305 (101.9363) | 276.502 (99.4242)
  Week 6: number analyzed (Participants) | 42 | 41 | 83 | 17 | 19 | 36
  Week 6 | 278.998 (178.6065) | 203.396 (122.0693) | 241.652 (157.0509) | 299.312 (118.7805) | 274.171 (128.5495) | 286.043 (122.9241)

7. Secondary Outcome: Biomarkers of Exposure - Total Nicotine Equivalents
Description: Total 24 hour urine will be collected to evaluate changes in total nicotine equivalents before, during, and after switching to VLN cigarettes. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: Summary of Urinary Tneq Mass Excreted (mg/24 hour) by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: mg/24 hour
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 21 | 20 | 41
mg/24 hour
  Week -1 | 17.511 (6.1103) | 15.885 (5.3291) | 16.690 (5.7580) | 17.732 (6.3013) | 15.928 (5.9611) | 16.852 (6.1291)
  Week 2: number analyzed (Participants) | 48 | 43 | 91 | 21 | 20 | 41
  Week 2 | 5.404 (4.5528) | 3.616 (3.5530) | 4.559 (4.1858) | 16.962 (6.2675) | 15.279 (4.7106) | 16.141 (5.5594)
  Week 6: number analyzed (Participants) | 42 | 41 | 83 | 17 | 19 | 36
  Week 6 | 9.150 (6.1240) | 6.800 (5.2118) | 7.989 (5.7792) | 17.530 (7.3994) | 14.418 (5.5176) | 15.888 (6.5703)

8. Secondary Outcome: Biomarkers of Exposure - Carboxyhemoglobin (COHb)
Description: Blood will be drawn to evaluate COHb before, during, and after switching to VLN cigarettes. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: Week -1, and at 2 and 6 weeks.
Population: Summary of Blood COHb (% Saturation) by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: % Saturation
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 50 | 50 | 100 | 22 | 20 | 42
% Saturation
  Week -1 | 6.20 (1.801) | 5.69 (1.526) | 5.95 (1.680) | 5.25 (1.294) | 5.41 (1.322) | 5.33 (1.294)
  Week 2: number analyzed (Participants) | 49 | 45 | 94 | 21 | 20 | 41
  Week 2 | 7.10 (2.794) | 5.55 (2.167) | 6.36 (2.618) | 5.40 (1.206) | 5.59 (2.060) | 5.49 (1.659)
  Week 6: number analyzed (Participants) | 43 | 42 | 85 | 19 | 20 | 39
  Week 6 | 5.97 (1.930) | 4.63 (1.898) | 5.31 (2.019) | 5.56 (1.323) | 4.61 (1.259) | 5.07 (1.361)

9. Secondary Outcome: Biomarkers of Exposure -Cotinine
Description: Blood will be drawn to evaluate cotinine levels before, during, and after switching to VLN cigarettes. The baseline data were collected for participants at Week -1, and Week -1 data are reported per pre-switch Arms/Group assignment.
Time Frame: Week -1, and at 2 and 6 weeks.
Population: Blood was drawn to evaluate cotinine levels before, during, and after switching to VLN cigarettes at Week -1, Week 2 and Week 6.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VLN Non-Mentholated | VLN Mentholated | UB Mentholated | UB Non-Mentholated
Number analyzed (Participants) | 50 | 50 | 70 | 72
ng/mL
  Week -1: number analyzed (Participants) | 0 | 0 | 70 | 72
  Week -1 |  |  | 242.0 (111.1681285) | 221.4 (85.32850957)
  Week 2: number analyzed (Participants) | 49 | 45 | 20 | 21
  Week 2 | 58.8 (58.5318519) | 58.7 (60.58382526) | 223.9 (100.5596713) | 195.8 (77.043868)
  Week 6: number analyzed (Participants) | 43 | 42 | 20 | 19
  Week 6 | 102.0 (76.3105523) | 110.1 (102.5119239) | 207.2 (81.7796209) | 187.7 (71.86818497)

10. Secondary Outcome: Nicotine Pharmacokinetics - Maximum Nicotine Concentration (C-Max)
Description: Blood samples will be drawn at -5, 2, 5, 7, 10, 12, 15, 20, 30, 45, 60, 90, 120, 150 and 180 minutes relative to the start of cigarette smoking a single cigarette for determination of C-max at weeks -1, 2 and 6. The baseline data were collected for participants at Week -1, and Week -1 data are reported per pre-switch Arms/Group assignment.
Time Frame: Week -1, and at 2 and 6 weeks.
Population: Plasma Nicotine Pharmacokinetic Parameters (Cmax) Following use of VLN Non-Mentholated, VLN Mentholated, UB Non-Mentholated, UB Mentholated Cigarettes (Pharmacokinetic Population from ITT).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VLN Non-Mentholated | VLN Mentholated | UB Non-Mentholated | UB Mentholated
Number analyzed (Participants) | 12 | 10 | 12 | 12
ng/mL
  Week -1: number analyzed (Participants) | 0 | 0 | 12 | 12
  Week -1 |  |  | 13.28 (5.9925) | 12.98 (5.3932)
  Week 2: number analyzed (Participants) | 12 | 10 | 0 | 0
  Week 2 | 0.3264 (0.15367) | 0.3561 (0.20204) |  |
  Week 6: number analyzed (Participants) | 12 | 10 | 0 | 0
  Week 6 | 0.4026 (0.15292) | 0.3259 (0.16294) |  |

11. Secondary Outcome: Nicotine Pharmacokinetics - Peak Nicotine Time (T-Max)
Description: Blood samples will be drawn at -5, 2, 5, 7, 10, 12, 15, 20, 30, 45, 60, 90, 120, 150 and 180 minutes relative to the start of cigarette smoking a single cigarette for determination of T-Max at weeks -1, 2 and 6. The baseline data were collected for participants at Week -1, and Week -1 data are reported per pre-switch Arms/Group assignment.
Time Frame: Week -1, and at 2 and 6 weeks.
Population: Plasma Nicotine Pharmacokinetic Parameters (Tmax) Following Use of VLN Non-Mentholated, VLN Mentholated, UB Mentholated and UB Non-Mentholated Cigarettes (Pharmacokinetic Population from ITT).
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | VLN Non-Mentholated | VLN Mentholated | UB Mentholated | UB Non-Mentholated
Number analyzed (Participants) | 12 | 10 | 12 | 12
hr
  Week -1: number analyzed (Participants) | 0 | 0 | 12 | 12
  Week -1 |  |  | 13.60 (5.2610) | 0.1408 (0.041525)
  Week 2: number analyzed (Participants) | 12 | 10 | 0 | 0
  Week 2 | 0.1154 (0.040675) | 0.1430 (0.063681) |  |
  Week 6: number analyzed (Participants) | 12 | 10 | 0 | 0
  Week 6 | 0.1446 (0.084195) | 0.2895 (0.43017) |  |

12. Secondary Outcome: Nicotine Pharmacokinetics - Area Under Nicotine Concentration Curve (AUC)
Description: Blood samples will be drawn at -5, 2, 5, 7, 10, 12, 15, 20, 30, 45, 60, 90, 120, 150 and 180 minutes relative to the start of cigarette smoking a single cigarette for determination of AUC at weeks -1, 2 and 6. The baseline data were collected for participants at Week -1, and Week -1 data are reported per pre-switch Arms/Group assignment.
Time Frame: Week -1, and at 2 and 6 weeks.
Population: Plasma Nicotine Pharmacokinetic Parameters (AUC0-180) Following Use of VLN Non-Mentholated, VLN Mentholated, UB Mentholated and UB Non-Mentholated Filtered Cigarettes (Pharmacokinetic Population from ITT).
Measure: Mean (Standard Deviation); unit: mg*hr/mL
Arm/Group | VLN Non-Mentholated | VLN Mentholated | UB Mentholated | UB Non-Mentholated
Number analyzed (Participants) | 12 | 10 | 12 | 12
mg*hr/mL
  Week -1: number analyzed (Participants) | 0 | 0 | 12 | 12
  Week -1 |  |  | 13.60 (5.2610) | 13.18 (4.0648)
  Week 2: number analyzed (Participants) | 12 | 10 | 0 | 0
  Week 2 | 0.2006 (0.19107) | 0.2264 (0.20588) |  |
  Week 6: number analyzed (Participants) | 12 | 10 | 0 | 0
  Week 6 | 0.2620 (0.15446) | 0.2348 (0.20330) |  |

13. Secondary Outcome: Smoking Topography - Puff Duration
Description: Puff duration will be measured before, during, and after switching to VLN cigarettes. Topography will be measured during an ad libitum smoking session. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: Summary of Puffing Topography Parameters by Study Product Group and Study Week (ITT Population). Puff topography was conducted in a randomly-selected subset of 18 non-menthol and 18 menthol cigarette smokers at a single site. The randomly-selected subjects have been assigned to switch to smoking very low nicotine (VLN) cigarettes.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined
Number analyzed (Participants) | 18 | 18 | 36
seconds
  Week -1 | 23.494 (7.9301) | 27.783 (7.6979) | 25.639 (8.0036)
  Week 2: number analyzed (Participants) | 16 | 17 | 33
  Week 2 | 23.282 (8.1071) | 24.559 (6.9773) | 23.940 (7.4545)
  Week 6: number analyzed (Participants) | 17 | 15 | 32
  Week 6 | 21.966 (7.0242) | 22.122 (6.4746) | 22.039 (6.6636)

14. Secondary Outcome: Smoking Topography - Puff Volume
Description: Puff volume will be measured before, during, and after switching to VLN cigarettes. Topography will be measured during an ad libitum smoking session. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined
Number analyzed (Participants) | 18 | 18 | 36
mL
  Week -1 | 50.7496 (12.88508) | 57.8934 (23.65244) | 54.3215 (19.11782)
  Week 2: number analyzed (Participants) | 16 | 17 | 33
  Week 2 | 44.6595 (13.48557) | 49.7368 (13.17315) | 47.2751 (13.36612)
  Week 6: number analyzed (Participants) | 17 | 15 | 32
  Week 6 | 47.9733 (13.25475) | 46.7513 (11.63150) | 47.4005 (12.33536)

15. Secondary Outcome: Smoking Topography - Peak Puff Flow Rate
Description: Peak Puff Flow Rate will be measured before, during, and after switching to VLN cigarettes. Topography will be measured during an ad libitum smoking session. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined
Number analyzed (Participants) | 18 | 18 | 36
mL/sec
  Week -1 | 44.3213 (10.85319) | 45.9639 (20.10163) | 45.1426 (15.94278)
  Week 2 | 39.7010 (13.72368) | 41.4412 (9.94555) | 40.5975 (11.76950)
  Week 6 | 43.4274 (14.75467) | 40.0195 (9.05336) | 41.8300 (12.34352)

16. Secondary Outcome: Smoking Topography - Average Flow Rate
Description: Average Puff Flow Rate will be measured before, during, and after switching to VLN cigarettes. Topography will be measured during an ad libitum smoking session. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined
Number analyzed (Participants) | 18 | 18 | 36
mL/sec
  Week -1 | 27.8305 (8.55885) | 28.5428 (12.99509) | 28.1866 (10.85056)
  Week 2: number analyzed (Participants) | 16 | 17 | 33
  Week 2 | 23.6309 (7.84344) | 25.4534 (5.68677) | 24.5698 (6.77219)
  Week 6: number analyzed (Participants) | 17 | 15 | 32
  Week 6 | 26.7164 (9.72496) | 24.1247 (5.15403) | 25.5016 (7.90798)

17. Secondary Outcome: Smoking Topography - Inter-puff Interval
Description: Inter-puff interval will be measured before, during, and after switching to VLN cigarettes. Topography will be measured during an ad libitum smoking session. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2 and 6 weeks.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined
Number analyzed (Participants) | 18 | 18 | 36
sec
  Week -1 | 30.269 (10.2050) | 29.222 (8.2654) | 29.746 (9.1677)
  Week 2: number analyzed (Participants) | 16 | 17 | 33
  Week 2 | 24.280 (9.2227) | 26.624 (12.1134) | 25.488 (10.7076)
  Week 6: number analyzed (Participants) | 17 | 15 | 32
  Week 6 | 21.044 (7.1810) | 27.215 (11.4332) | 23.937 (9.7693)

18. Secondary Outcome: Subjective Effects -Fagerstrom Test for Cigarette Dependance (FTCD)
Description: Subjects will answer a Fagerstrom Test for Cigarette Dependance (FTCD) questionnaire which contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence.The Fagerstrom Test for Nicotine Dependence, is scored from 0 to 1 for yes/no items and 0 to 3 for multiple-choice items.The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the greater the patient's physical dependence on nicotine. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2, 4, and 6 weeks.
Population: Summary of FTCD Score by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 20 | 22 | 42
score on a scale
  Week -1 | 5.2 (1.60) | 6.0 (1.53) | 5.6 (1.61) | 5.2 (1.46) | 5.4 (1.73) | 5.3 (1.59)
  Week 2: number analyzed (Participants) | 46 | 47 | 93 | 19 | 21 | 40
  Week 2 | 5.0 (1.79) | 6.3 (1.61) | 5.7 (1.81) | 5.2 (1.87) | 4.9 (1.92) | 5.1 (1.88)
  Week 4: number analyzed (Participants) | 41 | 43 | 84 | 20 | 19 | 39
  Week 4 | 4.8 (1.44) | 6.3 (1.71) | 5.6 (1.76) | 5.3 (2.02) | 5.3 (1.85) | 5.3 (1.92)
  Week 6: number analyzed (Participants) | 42 | 43 | 85 | 20 | 19 | 39
  Week 6 | 4.7 (1.65) | 6.0 (1.68) | 5.4 (1.78) | 5.4 (1.98) | 5.2 (2.04) | 5.3 (1.99)

19. Secondary Outcome: Subjective Effects -Brief Questionnaire of Smoking Urges (QSU-Brief)
Description: Subjects will answer a Brief Questionnaire of Smoking Urges (QSU-Brief). QSU is on a scale of 1-7, with 1 being strongly disagree and 7 being strongly agree. The average score of the following is taken to determine the Factor Score 1 and Factor Score 2; Factor 1: Average of Questions 1, 3, 6, 7, and 10; Factor 2: Average of Questions 2, 4, 5, 8, and 9. The score for each factor is calculated by summing the item scores; the total score is calculated by summing all questions together. The higher the score, the greater the urge to smoke. The total score range for this questionnaire is 10-70. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: Week -1, and at 2, 4, and 6 weeks.
Population: Summary of QSU-Brief Factor Score by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 20 | 22 | 42
score on a scale
  Week -1 | 4.2 (1.68) | 4.3 (1.70) | 4.3 (1.69) | 4.51 (1.50) | 3.8 (1.26) | 4.1 (1.41)
  Week 2: number analyzed (Participants) | 46 | 47 | 93 | 19 | 21 | 40
  Week 2 | 3.7 (1.87) | 5.4 (1.50) | 4.5 (1.88) | 4.3 (1.74) | 3.7 (1.48) | 4.0 (1.61)
  Week 4: number analyzed (Participants) | 41 | 43 | 84 | 20 | 19 | 39
  Week 4 | 3.8 (1.68) | 3.9 (1.47) | 3.8 (1.56) | 3.8 (1.47) | 3.7 (1.42) | 3.7 (1.43)
  Week 6: number analyzed (Participants) | 42 | 43 | 85 | 20 | 19 | 39
  Week 6 | 3.4 (1.70) | 4.4 (1.68) | 3.9 (1.75) | 4.1 (1.57) | 3.5 (1.57) | 3.8 (1.57)

20. Secondary Outcome: Subjective Effects - Minnesota Nicotine Withdrawal Scale - Revised (MNWS-R)
Description: Subjects will answer a MNWS-R questionnaire. The MNWS is considered as the briefest scale among the self-report measures of nicotine withdrawal symptoms currently available. The original MNWS was developed by Hughes and Hatsukami in 1986. It consisted of nine nicotine withdrawal symptoms including craving. The scale was modified to reflect changes made in the fourth edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for nicotine withdrawal. The total score of the scale range from 0 to 36 depending on participant's rate for the symptoms as not present (0), slight (1), mild (2), moderate (3), and severe (4). A high total score implies high nicotine addiction. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2, 4, and 6 weeks.
Population: Summary of MNWS-R Total Score by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 20 | 22 | 42
score on a scale
  Week -1 | 8.1 (7.56) | 13.0 (8.77) | 10.6 (8.52) | 10.6 (9.68) | 9.2 (7.49) | 9.9 (8.52)
  Week 2: number analyzed (Participants) | 46 | 47 | 93 | 19 | 21 | 40
  Week 2 | 8.4 (8.53) | 16.0 (9.74) | 12.3 (9.88) | 8.1 (9.02) | 9.0 (6.94) | 8.6 (7.90)
  Week 4: number analyzed (Participants) | 41 | 43 | 84 | 20 | 19 | 39
  Week 4 | 6.5 (7.67) | 13.5 (10.55) | 10.1 (9.86) | 8.4 (8.76) | 7.8 (7.10) | 8.1 (7.89)
  Week 6: number analyzed (Participants) | 42 | 43 | 85 | 20 | 19 | 39
  Week 6 | 5.4 (6.17) | 13.4 (10.01) | 9.5 (9.22) | 7.5 (7.32) | 8.3 (7.53) | 7.9 (7.33)

21. Secondary Outcome: Subjective Effects - Perceived Health Risks
Description: Subjects will answer a Perceived health risks questionnaire. The subjects indicated their perception of the risk of becoming addicted to the cigarette they were currently using on a scale from 1 to 10. Scale =1 was a very low risk of becoming addicted and Scale =10 was a very high risk of becoming addicted. The baseline data were collected for participants at Week -1, and Week -1 data are reported per post-switch Arms/Group randomization (instead of pre-switch Arms/Group assignment).
Time Frame: -1 week, and at 2, 4, and 6 weeks.
Population: Summary of Perceived Health Risk Scale by Study Product Group and Study Week (ITT Population)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VLN Non-Mentholated | VLN Mentholated | VLN Combined | UB Non-Mentholated | UB Mentholated | UB Combined
Number analyzed (Participants) | 49 | 50 | 99 | 20 | 22 | 42
units on a scale
  Week -1 | 7.0 (2.17) | 7.6 (2.04) | 7.3 (2.12) | 6.6 (2.09) | 7.7 (2.25) | 7.1 (2.23)
  Week 2: number analyzed (Participants) | 46 | 47 | 93 | 19 | 21 | 40
  Week 2 | 3.4 (2.73) | 4.0 (3.02) | 3.7 (2.88) | 6.8 (2.07) | 7.0 (2.68) | 6.9 (2.38)
  Week 4: number analyzed (Participants) | 41 | 43 | 84 | 20 | 19 | 39
  Week 4 | 3.4 (2.86) | 3.4 (2.55) | 34 (2.69) | 6.7 (2.37) | 7.4 (2.55) | 7.0 (2.45)
  Week 6: number analyzed (Participants) | 42 | 43 | 85 | 20 | 19 | 39
  Week 6 | 3.2 (2.89) | 3.6 (2.79) | 3.4 (2.83) | 6.6 (1.70) | 6.9 (2.54) | 6.7 (2.12)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after the start of Week 1 product use through follow-up call at Week 7.
Groups:
- Usual Brand Non-Metholated: Subjects will be switched from their usual brand to smoke Very Low Nicotine king size non-Menthol cigarettes
  Non-Menthol Very Low Nicotine Cigarettes: King size non-menthol cigarettes containing 0.4mg nicotine /g tobacco
- Usual Brand Metholated: Subjects will be switched from their usual brand to smoke Very Low Nicotine king size cigarettes
  Menthol Very Low Nicotine Cigarettes: King size menthol cigarettes containing 0.4mg nicotine /g tobacco
Arm/Group | Non-Menthol Very Low Nicotine Cigarettes | Menthol Very Low Nicotine Cigarettes | Usual Brand Non-Metholated | Usual Brand Metholated
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/50 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 11/50 | 11/50 | 5/22 | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Menthol Very Low Nicotine Cigarettes (N=50) | Menthol Very Low Nicotine Cigarettes (N=50) | Usual Brand Non-Metholated (N=22) | Usual Brand Metholated (N=20)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Menthol Very Low Nicotine Cigarettes (N=50) | Menthol Very Low Nicotine Cigarettes (N=50) | Usual Brand Non-Metholated (N=22) | Usual Brand Metholated (N=20)
Headache (Nervous system disorders) | 8 | 6 | 5 | 3
Irritability (Psychiatric disorders) | 3 | 5 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03571724/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT03571724/SAP_001.pdf